CLINICAL TRIAL: NCT01562925
Title: Randomized Controlled Study for Evaluation of the Impact of Red Wine, White Wine and Beer Intake on Contrast-Medium Induced Acute Kidney Injury
Brief Title: Effect of Red Wine, White Wine and Beer on Contrast-Medium Induced Acute Kidney Injury
Acronym: RenPro-II-WINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Fikret Er, MD, Assistant Professor, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RenPro-WINE
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Renal Failure/ Kidney Disease; Contrast-medium Induced Acute Kidney Injury
MeSH Terms: interventions — Beer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Red Wine (Active Comparator): Patients assigned to red wine group will receive standard care plus two doses of red wine: the evening before contrast-medium use and the morning of contrast-medium exposure
  Interventions: Dietary Supplement: Red wine
- White wine (Active Comparator)
  Interventions: Dietary Supplement: White wine
- Beer (Active Comparator)
  Interventions: Dietary Supplement: Beer
- Control (No Intervention): Patients assigned to control group will receive standard care. Patients receive ordinary still water without alcohol the evening before(7.8 ml per kg bodyweight) and 60-120 minutes before contrast exposure (at least 3.9 ml per kg bodyweight)

INTERVENTIONS:
Dietary Supplement: Red wine — Red wine First dosage: 3 ml per kg bodyweight (the evening before contrast medium exposure) Second dosage: 1.5 ml per kg bodyweight (60-120 minutes before contrast medium exposure
  Other Names: Frühburgunder 2006, Spätlese Trocken, Schloss Westerhaus, Rheinhessen, 12.5% vol
  Arms: Red Wine
Dietary Supplement: White wine — White wine First dosage: 3.3 ml per kg bodyweight (the evening before contrast medium exposure) Second dosage: 1.7 ml per kg bodyweight (60-120 minutes before contrast medium exposure
  Other Names: Riesling feinherb 2009, Dr. Willkomm, Bernkastel-Kues, 12.5% vol
  Arms: White wine
Dietary Supplement: Beer — Beer First dosage: 7.8 ml per kg bodyweight (the evening before contrast medium exposure) Second dosage: 3.9 ml per kg bodyweight (60-120 minutes before contrast medium exposure
  Other Names: Cologne mild beer (Kölsch); Gaffel Kölsch, Gaffel Brauerei Cologne, 4.8% vol
  Arms: Beer

SUMMARY:
Patients with impaired renal function are at elevated risk for development of contrast-medium induced acute kidney injury (CI-AKI). CI-AKI is associated with increased risk for cardiovascular morbidity and mortality. Effective CI-AKI prevention strategies are needed.

The RenPro-II-WINE Trial was designed to test the hypothesis whether moderate red wine consumption prior to contrast-medium use is effective in CI-AKI prevention.

Consecutive patients with impaired renal function undergoing elective coronary angiography will be assigned in one of four treatment arms: a. control patients receiving standard care b. patients receiving standard care plus red wine c. patients receiving standard care plus white wine d. patients receiving standard care plus beer This study will give important answers on how to prevent CI-AKI in patients with impaired renal function undergoing contrast media exposure.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* impaired renal function (baseline estimated glomerular filtration rate of <60 ml/min)
* at least three of following comorbidities: hypertension, diabetes mellitus without insulin therapy, heart failure NYHA III and/or left ventricular ejection fraction <35%, peripheral artery disease, coronary artery disease

Exclusion Criteria:

* known alcohol addiction
* severe renal impairment (estimated glomerular filtration rate <15 ml/min and/or in chronic dialysis program
* Recent (<=30 days) contrast media exposure
* insulin therapy
* Patients enrolled in concomitant studies
* fertile women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
CI-AKI incidence | <48 hours after contrast-medium exposure
  Increment of serum-creatinin of 0.5 mg/dl or of at least 25% in 48 hours after contrast medium intake from baseline.

SECONDARY OUTCOMES:
Biomarkers assessing acute kidney injury | <48 hours
  Changes of urinary neutrophil gelatinase-associated lipocalin (NGAL), serum creatinin and cystatine after coronary angiogram.

CONTACTS AND LOCATIONS:
Locations (1):
- Herzzentrum der Universität zu Köln, Cologne, Germany

REFERENCES:
- See also: study group homepage — http://www.cardiovascular-research.org